CLINICAL TRIAL: NCT00859560
Title: Retrospective Survey of Bone Fracture in Post-Menopausal Breast Cancer Patients With Arimidex 1 mg as Adjuvant Therapy
Brief Title: Retrospective Survey of Bone Fracture in Patients With Arimidex 1mg
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Alain Huvenne, Senior Medical Marketing Director, AstraZeneca KK
Other Study IDs: NIS-OJP-ARI-2007/1
Record Dates: First submitted 2009-03-10; First posted 2009-03-11 (Estimated); Last update posted 2009-03-11 (Estimated); Status verified 2009-03

CONDITIONS: Breast Cancer
Keywords: Breast cancer; post-menopausal women; Arimidex; bone fracture
MeSH Terms: conditions — Breast Neoplasms; Fractures, Bone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

SUMMARY:
The retrospective survey is to investigate the incidence of bone fracture in post-menopausal breast cancer patients with Arimidex 1mg, who were previously registered for the clinical experience investigation.

ELIGIBILITY:
Inclusion Criteria:

* Post-menopausal breast cancer patients treated with Arimidex 1mg at the time of previously conducted clinical experience investigation.

Exclusion Criteria:

-

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Post-menoposal breast cancer patients who were previousely registered in clinical experience investigation with Arimidex 1mg as adjuvant therapy.
Sampling Method: Non-Probability Sample
Enrollment: 2205 (Actual)
Dates: Start 2008-01; Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Bone fracture incidence | Time since starting Arimidex

SECONDARY OUTCOMES:
Survival | Time since starting Arimidex
Bone density measurement | Time since starting Arimidex

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Japan Medical Director MD, Study Director — AstraZeneca